CLINICAL TRIAL: NCT01150279
Title: Simplifying Medical Abortion Provision: Exploring the Role of At-home Semi-Quantitative Pregnancy Tests for Medical Abortion Follow-up
Brief Title: Exploring the Role of At-home Semi-Quantitative Pregnancy Tests for Medical Abortion Follow-up
Status: Completed | Type: Observational
Sponsor: Gynuity Health Projects (Other)
Collaborators: Stanford University (Other); Secretaría de Salud del Distrito Federal (Unknown); Office National de la Famille et de la Population, Tunisia (Unknown); Maternité de la Rabta, Tunisia (Unknown); Clinique du Parc, Tunisia (Unknown)
Responsible Party: Sponsor
Other Study IDs: 6.1.3
Record Dates: First submitted 2010-05-13; First posted 2010-06-24 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Medical Abortion
Keywords: medical abortion; Medical Abortion Follow Up Care

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
This study will examine the feasibility, acceptability and usability of a semi-quantitative urine pregnancy test (dBest One Step hCG Panel Test Kit) for at-home follow-up after early medical abortion using mifepristone+misoprostol. The study seeks to:

1. Assess the feasibility of using this test in lieu of standard one-week clinic-based follow up for determination of complete abortion status as part of normal service delivery. In Mexico, follow up will be in two weeks, as is standard care in that .
2. To determine if women using this test at home understand how to use it and can correctly interpret the results; is it practical.
3. Assess women's and provider's acceptability of using at-home pregnancy tests in lieu of clinic-based follow up for confirmation of complete medical abortion in the future.

ELIGIBILITY:
Inclusion Criteria:

* Women age greater than or equal to 18 years
* Gestational age less than or equal to 63 days by last menstrual period (LMP), ultrasound or clinical assessment
* Agrees to return for follow-up visit and willing to provide an address and/or telephone number for purposes of follow-up
* Able to consent to study participation.

Inclusion Criteria for Mexico:

* Gestational age <_ 70 days from LMP
* Eligible for mifepristone- misoprostol medical abortion according to clinic guidelines
* Willing to follow instructions of the provider regarding use of the at-home pregnancy test
* Agrees to provide test results by phone to study coordinator on morning of schedule follow-up visit
* Willing to provide an address and/or telephone number for purposes of follow-up
* Agrees to return for standard follow-up visit
* Wishes to participate in the study
* Having easy access to a telephone and transportation
* Able to consent to study participation

Exclusion Criteria:

* Women less than 18 years of age
* Women not eligible for medical abortion services
* Women unable to provide contact information
* Women unable to sign the consent form

Exclusion Criteria for Mexico:

* Women not eligible for medical abortion services
* Women unable to provide contact information
* Women unable to sign the consent form

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women presenting to clinic seeking medical abortion
Sampling Method: Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2009-08; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Percent of women who correctly interpreted their results (in U.S. and Vietnam only) | 18 months

SECONDARY OUTCOMES:
Percent of women who felt confident in using the test and would be willing to use it in place of clinic-based follow up in the future | 18 months
The proportion of times the provider believes that each participant correctly read her test result | 18 months
Percent of providers who were comfortable with the urine pregnancy test determining whether women need to return or not for clinic-based follow-up | 18 months
The proportion of times that the semi-quantitative test correctly identifies all on going pregnancies | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul D Blumenthal, MD, MPH, Principal Investigator — Stanford University; Beverly Winikoff, MD, MPH, Principal Investigator — Gynuity Health Projects; Jennifer Blum, MPH, Principal Investigator — Gynuity Health Investigator; Patricio Sanhueza Smith, MD, Principal Investigator — Secretaría de Salud del Distrito Federal; Rym Fayala, MD, Principal Investigator — Office National de la Famille et de la Population; Ezzedine Sfar, Principal Investigator — Maternité de la Rabta; Hella Chelli, Principal Investigator — Clinique du Parc; Rasha Dabash, MPH, Study Director — Gynuity Health Projects
Locations (11):
- United States (4):
  - Stanford University Hospital, Palo Alto, California
  - Planned Parenthood Mar Monte, Sacramento, California
  - Family Planning Associates Group - Washington, Chicago, Illinois
  - Family Planning Associates- Elston, Chicago, Illinois
- Hospital Materno Infantil Nicolas M. Cedillo, Mexico City, Mexico
- Tunisia (5):
  - ONFP Ben Arous, Ben Arous
  - ONFP Nabeul, Nabeul
  - ONFP Sousse, Sousse
  - Clinique du Parc, Tunis
  - Maternite de la Rabta, Tunis
- HocMon District Hospital, Ho Chi Minh City, Vietnam

REFERENCES:
- [Derived] Dabash R, Shochet T, Hajri S, Chelli H, Hassairi AE, Haleb D, Labassi H, Sfar E, Temimi F, Koenig L, Winikoff B. Self-administered multi-level pregnancy tests in simplified follow-up of medical abortion in Tunisia. BMC Womens Health. 2016 Jul 30;16:49. doi: 10.1186/s12905-016-0327-1. PMID 27475998
- [Derived] Lynd K, Blum J, Ngoc NT, Shochet T, Blumenthal PD, Winikoff B. Simplified medical abortion using a semi-quantitative pregnancy test for home-based follow-up. Int J Gynaecol Obstet. 2013 May;121(2):144-8. doi: 10.1016/j.ijgo.2012.11.022. Epub 2013 Mar 7. PMID 23477704